CLINICAL TRIAL: NCT03870022
Title: Pivot Breath Sensor Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Marler, MD (Industry)
Collaborators: UserWise, LLC (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Marler, MD, Senior Director, Clinical and Medical Affairs, Pivot Health Technologies Inc.
Organization: Pivot Health Technologies Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C-150
Record Dates: First submitted 2019-03-05; First posted 2019-03-11 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Smoking Cessation; Smoking, Tobacco
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 18-80 years of age (Other): Single day study collecting 1 paired breath sample from each subject using two non-invasive breath sampling devices, as well as collecting participant responses to user documentation questions and rating scales.
  Interventions: Device: Pivot Breath Sensor System; Device: Similar Carbon Monoxide breath sensor system

INTERVENTIONS:
Device: Pivot Breath Sensor System — Collect breath sample from the Pivot Breath Sensor to measure the carbon monoxide in the participant's exhaled breath, along with recording responses to user documentation questions and rating scales.
Device: Similar Carbon Monoxide breath sensor system — Collect breath sample from a similar breath sensor to measure the carbon monoxide in the participant's exhaled breath.

SUMMARY:
A clinical study enrolling 70 subjects to:

* evaluate the user performance of the Pivot Breath Sensor
* compare measurements from the Pivot Breath Sensor to a similar device
* assess user documentation comprehension
* obtain feedback on the Pivot Breath Sensor via rating scales. No medical decisions will be made related to test results.

DETAILED DESCRIPTION:
The objectives of this performance study are to:

* Non-invasively measure carbon monoxide (CO) levels in the exhaled breath of study subjects using two different types of measurement devices.
* We will assess the correlation between the measured CO levels (in parts per million, or ppm) of the study CO breath sensor (Carrot Inc.) and a similar device.
* assess user documentation comprehension
* obtain feedback on the Pivot Breath Sensor via rating scales.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Owns and uses a smartphone
* Willing to sign the Informed Consent Form
* Resident of the United States
* Able to read and comprehend English

Exclusion Criteria:

* Prior experience with a study sponsored by Carrot Inc.
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jen Marler, Principal Investigator — Pivot Health Technologies Inc.
Locations (1):
- Carrot Inc., Redwood City, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 18-80 Year Old Smokers: Smokers aged 18-80 - collection of 1 paired breath sample from each subject using two non-invasive breath sampling devices, as well as collecting participant responses to user documentation questions and rating scales.
  Pivot Breath Sensor System: Collect breath sample from the Pivot Breath Sensor to measure the carbon monoxide in the participant's exhaled breath, along with recording responses to user documentation questions and rating scales.
  Bedfont - Micro+™ Smokerlyzer®: Bedfont - Micro+™ Smokerlyzer® : Predicate Device to measure carbon monoxide levels in one's breath..
Period: Overall Study
Arm/Group | 18-80 Year Old Smokers
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 18-80 Year Old Smokers
Number analyzed (Participants) | 70
Age, Customized [Count of Participants; unit: Participants]
  Age 18-49 | 34
  Age 50-80 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 44
  Hispanic, Latino, or Spanish Origin | 6
  Black or African American | 10
  Asian | 8
  American Indian or Alaska Native | 1
  Hawaiian or other Pacific Islander | 1
Region of Enrollment [Number; unit: participants]
  United States | 70
years smoking [Mean (Standard Deviation); unit: years] | 29.8 (14.8)

OUTCOME MEASURES:

1. Primary Outcome: User Performance of Pivot Breath Sensor
Description: Assess user performance of the study device at a single visit. Participants will be observed if they can set up the Pivot Breath Sensor, and whether they can use the device. Observer ratings include 'Successful' and 'Unsuccessful'. Specific attention will be given to assess if any harms can occur from observed use errors.
  "Successful" = the participant was able to complete the task independently, safely, effectively, and without difficulty.
  "Unsuccessful" = the participant was unable to complete the task independently, safely, effectively, and/or without difficulty. Includes instances where the participant required study moderator assistance.
Time Frame: Each study session lasted up to 60 minutes per participant. Use performance was assessed at approximately 10-15 minutes into the study session.
Measure: Count of Participants; unit: Participants
Arm/Group | 18-80 Year Old Smokers
Number analyzed (Participants) | 70
Participants
  Self-training: Successful | 68
  Self-training: Unsuccessful | 2
  Performance breath sample use and/or with use of reference materials: Successful | 70
  Performance breath sample use and/or with use of reference materials: Unsuccessful | 0

2. Primary Outcome: Compare Performance of Pivot Breath Sensor With a Similar Device.
Description: Compare study device performance with a similar device at a single visit.
  Participants will then be asked to use a similar CO breath sensor device. The correlation between the measured CO levels (in parts per million, or ppm) of the study CO breath sensor (Carrot Sense) and the similar breath sensor will be assessed.
Time Frame: Each study session lasted up to 60 minutes per participant.
Measure: Number; unit: Correlation coefficient (R-value)
Arm/Group | 18-80 Years of Age
Number analyzed (Participants) | 70
Correlation coefficient (R-value) | 0.9710

3. Secondary Outcome: User Documentation Assessment With Observer Ratings
Description: Participant understanding of user documentation will be assessed at single visit through interpretation of three different CO test results: green, orange, and red. User documentation used for the interpretation of each result includes: packaging information, quick start guide and user manual. Observer ratings include 'Successful' and 'Unsuccessful'.
  "Successful" = the participant was able to complete the task independently, safely, effectively, and without difficulty.
  "Unsuccessful" = the participant was unable to complete the task independently, safely, effectively, and/or without difficulty. Includes instances where the participant required study moderator assistance.
  Participant will be asked to assess the user documentation throughout the study session and will take approximately 10 minutes.
Time Frame: Each study session lasted up to 60 minutes per participant. The user documentation assessment with observer ratings was done between approximately 10 and 35 minutes into the study session.
Measure: Count of Participants; unit: Participants
Arm/Group | 18-80 Year Old Smokers
Number analyzed (Participants) | 70
Participants
  Interpretation of Green CO category after using reference materials: Successful | 69
  Interpretation of Green CO category after using reference materials: Unsuccessful | 1
  Interpretation of Orange CO category after using reference materials: Successful | 57
  Interpretation of Orange CO category after using reference materials: Unsuccessful | 13
  Interpretation of Red CO category after using reference materials: Successful | 70
  Interpretation of Red CO category after using reference materials: Unsuccessful | 0

4. Secondary Outcome: Participant Feedback Using Rating Scale
Description: Participant will be asked to provide ratings on the following:
  * How would you rate the ease or difficulty using the device?
  * How clear or unclear was the Quick Start Guide? Why?
  * How clear or unclear was the Packaging? Why?
  * How clear or unclear was the User Manual on the iPad? Why?
  * Overall, how clear or unclear were the provided reference materials? Why?
  * How easy or difficult was it to understand and interpret the test results? Why?
  The participant will use the following rating scale:
  5 - Very Easy 4 - Easy 3 - Neither Easy nor Difficult 2 - Difficult
  1 - Very Difficult Not Applicable
  Participant will provide the ratings prior to the conclusion of the study session. Participant assessment with questionnaire rating scales will take approximately 1-2 minutes each.
Time Frame: Each study session lasted up to 60 minutes per participant. Use performance was assessed with rating scales at approximately 35 minutes into the study session.
Measure: Count of Participants; unit: Participants
Arm/Group | 18-80 Year Old Smokers
Number analyzed (Participants) | 70
Participants
  How would you rate the ease or difficulty using the device?: Very Easy | 27
  How would you rate the ease or difficulty using the device?: Easy | 32
  How would you rate the ease or difficulty using the device?: Neither Easy nor Difficult | 9
  How would you rate the ease or difficulty using the device?: Difficult | 2
  How would you rate the ease or difficulty using the device?: Very Difficult | 0
  How would you rate the ease or difficulty using the device?: Not Applicable | 0
  How clear or unclear was the Quick Start Guide? Why?: Very Easy | 42
  How clear or unclear was the Quick Start Guide? Why?: Easy | 16
  How clear or unclear was the Quick Start Guide? Why?: Neither Easy nor Difficult | 6
  How clear or unclear was the Quick Start Guide? Why?: Difficult | 1
  How clear or unclear was the Quick Start Guide? Why?: Very Difficult | 0
  How clear or unclear was the Quick Start Guide? Why?: Not Applicable | 5
  How clear or unclear was the Packaging? Why?: Very Easy | 54
  How clear or unclear was the Packaging? Why?: Easy | 12
  How clear or unclear was the Packaging? Why?: Neither Easy nor Difficult | 3
  How clear or unclear was the Packaging? Why?: Difficult | 1
  How clear or unclear was the Packaging? Why?: Very Difficult | 0
  How clear or unclear was the Packaging? Why?: Not Applicable | 0
  How clear or unclear was the User Manual on the iPad? Why?: Very Easy | 11
  How clear or unclear was the User Manual on the iPad? Why?: Easy | 8
  How clear or unclear was the User Manual on the iPad? Why?: Neither Easy nor Difficult | 2
  How clear or unclear was the User Manual on the iPad? Why?: Difficult | 2
  How clear or unclear was the User Manual on the iPad? Why?: Very Difficult | 1
  How clear or unclear was the User Manual on the iPad? Why?: Not Applicable | 46
  Overall, how clear or unclear were the provided reference materials? Why?: Very Easy | 39
  Overall, how clear or unclear were the provided reference materials? Why?: Easy | 27
  Overall, how clear or unclear were the provided reference materials? Why?: Neither Easy nor Difficult | 3
  Overall, how clear or unclear were the provided reference materials? Why?: Difficult | 1
  Overall, how clear or unclear were the provided reference materials? Why?: Very Difficult | 0
  Overall, how clear or unclear were the provided reference materials? Why?: Not Applicable | 0
  How easy or difficult was it to understand and interpret the test results? Why?: Very Easy | 48
  How easy or difficult was it to understand and interpret the test results? Why?: Easy | 16
  How easy or difficult was it to understand and interpret the test results? Why?: Neither Easy nor Difficult | 3
  How easy or difficult was it to understand and interpret the test results? Why?: Difficult | 2
  How easy or difficult was it to understand and interpret the test results? Why?: Very Difficult | 1
  How easy or difficult was it to understand and interpret the test results? Why?: Not Applicable | 0

ADVERSE EVENTS:
Time Frame: Adverse events were observed for over the 60-minute long study session for each participant.
Arm/Group | 18-80 Year Old Smokers
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT03870022/Prot_SAP_001.pdf